CLINICAL TRIAL: NCT04363294
Title: Targeted Testing for Transthyretin Cardiac Amyloid Among Aortic Stenosis Patients-Pilot
Brief Title: Targeted Testing for ATTR Among Aortic Stenosis Patients-Pilot
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: grant was not approved, no subjects enrolled
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Mid America Heart Institute (Other)
Responsible Party: Principal Investigator, Anthony Bavry, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: STU-2020-0386
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Aortic Valve Stenosis; Cardiac Amyloidosis
Keywords: aortic stenosis; transthyretin cardiac amyloid; transcatheter aortic valve replacement; AortoVentricular index; ATTR; TAVR; AVi; invasive cardiac hemodynamics
MeSH Terms: conditions — Aortic Valve Stenosis; Amyloid Neuropathies, Familial

STUDY DESIGN:
Intervention Model Description: Participants undergoing TAVR for symptomatic severe aortic stenosis, with pre-TAVR echocardiography and post-implantation invasive hemodynamic assessment are eligible for study participation. The AVi will be recorded from post-implantation invasive hemodynamic assessment. Participants will undergo bone scintigraphy (99mTc-pyrophosphate Planar/SPECT imaging) within 28 days after TAVR. Participants with abnormal bone scintigraphy require evaluation for a monoclonal protein with blood/urine laboratory testing, and possible tissue biopsy/Hematology consultation to exclude light-chain amyloidosis. Participants who are ATTR positive will receive comprehensive heart failure management and possible genetic testing to evaluate for mutated ATTR.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Other): Patients who had TAVR and underwent evaluation for ATTR with PYP scan
  Interventions: Diagnostic Test: PYP scan

INTERVENTIONS:
Diagnostic Test: PYP scan — 99mTc-labeled pyrophosphate
  Other Names: Bone scan

SUMMARY:
Our ultimate goal is to design a multi-center randomized trial to test the hypothesis that targeted testing for transthyretin cardiac amyloid (ATTR) will improve survival and health status among aortic stenosis patients who undergo transcatheter aortic valve replacement (TAVR). The hypothesis of this pilot study is to evaluate if invasive cardiac hemodynamics obtained after TAVR, by using the AortoVentricular index (AVi), can be used as a novel test to help identify participants with ATTR.

Aim 1. To determine if an abnormal AVi value can identify ATTR among aortic stenosis patients undergoing TAVR.

Aim 2. To determine if s' from echocardiography plus AVi can enhance the prediction of ATTR among aortic stenosis patients undergoing TAVR.

Aim 3. To design a pilot trial to improve patient outcomes after TAVR by targeted testing for ATTR.

DETAILED DESCRIPTION:
Aim 1. To determine if an abnormal AVi value can identify ATTR among aortic stenosis patients undergoing TAVR. Patients undergoing TAVR for symptomatic severe aortic stenosis, with pre-TAVR echocardiography and post-implantation invasive hemodynamic assessment are eligible for study participation. The AVi will be recorded from post-implantation invasive hemodynamic assessment. Participants will undergo bone scintigraphy (99mTc-pyrophosphate Planar/SPECT imaging) within 28 days after TAVR. Participants with abnormal bone scintigraphy require evaluation for a monoclonal protein with blood/urine laboratory testing, and possible tissue biopsy/Hematology consultation to exclude light-chain amyloidosis. Participants who are ATTR positive will receive comprehensive heart failure management and possible genetic testing to evaluate for mutated ATTR. The prevalence of ATTR will be reported among participants with AVi <0.5 versus ≥0.5 mm Hg/beats per minute. Test performance of AVi to predict ATTR will be reported.

Aim 2. To determine if s' obtained from echocardiography tissue Doppler imaging plus AVi can enhance the prediction of ATTR among aortic stenosis patients undergoing TAVR. The s' will be recorded from pre-TAVR tissue Doppler imaging of the mitral annulus. The prevalence of ATTR will be reported among participants with both s' ≤6 cm/second and AVi <0.5 mm Hg/beats per minute versus s' >6 cm/second and AVi <0.5 mm Hg/beats per minute.

Aim 3. To design a pilot trial to improve patient outcomes after TAVR by targeted testing for ATTR. The change in Kansas City Cardiomyopathy Questionnaire-12 from baseline to 12-months and survival with reasonable quality of life at 12-months will be reported among participants who are ATTR positive vs. ATTR negative.

ELIGIBILITY:
Inclusion Criteria:

* Successful implantation of a transcatheter heart valve with a commercially available valve (i.e. Sapien 3, Sapien Ultra, Evolut R, Evolut Pro, Evolut Pro+, or Lotus Edge) for native or bioprosthetic aortic stenosis
* Pre-implantation echocardiography with tissue Doppler imaging, if feasible
* Post-implantation invasive cardiac hemodynamics

Exclusion Criteria:

* Age <75 years
* Moderate to severe paravalvular aortic regurgitation on post-operative echocardiography

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Prevalence ATTR with AVi <0.5 | Within 28 days after TAVR when bone scan completed
  Prevalence of ATTR among participants with AVi <0.5 mm Hg/beats per minute
Prevalence ATTR with AVi ≥0.5 | Within 28 days after TAVR when bone scan completed
  Prevalence of ATTR among participants with AVi ≥0.5 mm Hg/beats per minute

SECONDARY OUTCOMES:
Sensitivity AVi | Within 28 days after TAVR when bone scan completed
  Sensitivity of AVi <0.5 mm Hg/beats per minute
Specificity AVi | Within 28 days after TAVR when bone scan completed
  Specificity of AVi ≥0.5 mm Hg/beats per minute
Positive predictive value AVi | Within 28 days after TAVR when bone scan completed
  Positive predictive value of AVi <0.5 at predicting ATTR
Negative predictive value AVi | Within 28 days after TAVR when bone scan completed
  Negative predictive value of AVi ≥0.5 at ruling out ATTR

OTHER OUTCOMES:
Prevalence ATTR with s'<6 plus AVi <0.5 | Within 28 days after TAVR when bone scan completed
  Prevalence of ATTR among participants with both s'<6 and AVi <0.5 mm Hg/beats per minute
Prevalence ATTR with s'≥6 plus AVi <0.5 | Within 28 days after TAVR when bone scan completed
  Prevalence of ATTR among participants with both s'≥6 and AVi <0.5 mm Hg/beats per minute
KCCQ-12 | 1 year after TAVR
  Kansas City Cardiomyopathy Questionnaire(KCCQ) - a shortened 12 question version of the 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Favorable outcome | 1 year after TAVR
  Proportion of subjects who are alive with reasonable quality of life. Reasonable quality of life is defined as KCCQ-12 ≥60 without any meaningful worsening (decrease in KCCQ-12 summary score ≥10).

CONTACTS AND LOCATIONS:
Overall Officials: Anthony A Bavry, MD MPH, Principal Investigator — University of Texas Southwestern Medical Center

IPD SHARING:
Plan to Share IPD: Yes
The primary investigator will upload de-identified individual data after study results have been published
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available after study results have been published
Access Criteria: The primary investigator will upload study protocol, statistical analysis plan, informed consent form, and clinical study report after study results have been published